CLINICAL TRIAL: NCT01665950
Title: Simvastatin Augmentation of Lithium Treatment in Bipolar Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Roy Perlis, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011P002545
Record Dates: First submitted 2012-04-09; First posted 2012-08-16 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Simvastatin-Simvastatin (Experimental): Subjects will receive simvastatin in phase 1 (4 weeks) and phase 2 (4 weeks)
  Interventions: Drug: Simvastatin
- Placebo->Simvastatin (Experimental): Placebo non-responders after the 1st 4 weeks will be re-randomized 1:1 to placebo or simvastatin for the next 4 weeks
  Interventions: Drug: Simvastatin; Drug: Placebo
- Placebo-Placebo (Placebo Comparator): Placebo nonresponders for the 1st 4 weeks will be re-randomized 1:1 to placebo or simvastatin for the subsequent 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — The study uses the Sequential Parallel Comparison design (SPCD), with two 4-week phases: n=30 subjects are randomized 1:1 to simvastatin versus placebo add-on for 4 weeks, with the nonresponders re-randomized 1:1 for a further 4 weeks. The SPCD will allow us to pool data from both phases to estimate the simvastatin treatment effect. Subjects who respond in phase 1, and all subjects who receive simvastatin in phase 1, continue blinded treatment in phase 2 to preserve the blind, but only phase 1 results are analyzed. Dosage for simvastatin or matched placebo 20mg daily for 8 weeks.
  Arms: Placebo->Simvastatin; Simvastatin-Simvastatin
Drug: Placebo — Subjects (n=15) are randomized to placebo add-on for 4 weeks, with the nonresponders re-randomized 1:1 to statin vs placebo for a further 4 weeks. Subjects who respond in phase 1 continue blinded treatment in phase 2 to preserve the blind, but only phase 1 results are analyzed. Dosage for simvastatin or matched placebo 20mg daily for 8 weeks.
  Arms: Placebo->Simvastatin; Placebo-Placebo

SUMMARY:
Primary Aim: To estimate the antidepressant efficacy of simvastatin versus placebo as an adjunct to lithium, valproate, and/or other atypical antipsychotic therapy among individuals with bipolar I disorder in a nonpsychotic major depressive episode.

Hypothesis: Simvastatin will be superior to placebo in improvement of depressive symptoms assessed by the Montgomery-Asberg Depression Rating Scale (MADRS).

DETAILED DESCRIPTION:
(see brief summary)

ELIGIBILITY:
Inclusion:

* Age 18-65
* written informed consent
* meets Diagnostic and Statistical Manual - IV (DSM-IV) criteria (by Structured Clinical Interview for DSM-IV (SCID-I/P)) for bipolar I disorder, current episode depressed
* Montgomery-Asberg Depression Scale (MADRS) score of at least 20 (i.e., moderate depression) and no greater than 34 (i.e., severe depression) at screen and baseline visit
* Young Mania Rating Scale (YMRS) score < 12 at screen and baseline visit
* currently treated with a lithium preparation (carbonate or citrate) at stable dose for at least 4 wks with level >0.4 and <1.0; and/or valproate at stable dose for at least 4 wks at level >60 and <110; and/or other atypical antipsychotic at stable dose for at least 4 weeks (at least minimum FDA-labeled dose).

Exclusion:

* Psychotic features in the current episode, as assessed by YMRS item #8>6
* felt by the study clinician to require inpatient hospitalization for adequate management
* more than 3 failed pharmacologic interventions in the current major depressive episode, exclusive of primary mood stabilizer
* current substance use disorder other than nicotine, by SCID-I/P
* pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy)
* women who are breastfeeding
* serious suicide or homicide risk, as assessed by evaluating clinician
* other unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease, based on review of medical history, physical examination, and screening laboratory tests
* patients who have taken an investigational psychotropic drug within the last 30 days
* patients receiving additional anticonvulsant, antipsychotic, or antidepressant within 1 week prior to study entry
* patients requiring continued treatment with excluded medications (see below).

Excluded medications: other statins, which could influence Wnt signaling; any other drug known to interact with simvastatin, including potent inhibitors/inducers of CYP3A4 such as itraconazole, ketoconazole, posaconazole, erythromycin, clarithromycin, telithromycin, voriconazole, cyclosporine or danazol; gemfibrozil or other lipid-lowering drugs that can cause myopathy when given alone; amiodarone, ranolazine, verapamil, diltiazem, or amlodipine; niacin; digoxin; coumarin anticoagulants; colchicine; nefazodone; protease inhibitors including ritonavir, indinavir, nelfinavir, or saquinavir.

Allowed: benzodiazepines and sedative-hypnotic agents if dosage has been stable for 2 weeks prior to study entry; thyroid or estrogen replacement provided dosage has been stable for 1 month; antidepressants, antipsychotics, and anticonvulsants provided dosage has been stable for 1 week prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy H Perlis, MD, MSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin-Simvastatin: Subjects will receive simvastatin in phase 1 (4 weeks) and phase 2 (4 weeks)
  Simvastatin: The study uses the Sequential Parallel Comparison design (SPCD), with two 4-week phases: Subjects are randomized 1:1 to simvastatin versus placebo add-on for 4 weeks, with the nonresponders re-randomized 1:1 for a further 4 weeks. The SPCD will allow us to pool data from both phases to estimate the simvastatin treatment effect. Subjects who respond in phase 1, and all subjects who receive simvastatin in phase 1, continue blinded treatment in phase 2 to preserve the blind, but only phase 1 results are analyzed. Dosage for simvastatin or matched placebo 20mg daily for 8 weeks.
- Placebo->Simvastatin: Placebo non-responders after the 1st 4 weeks will be re-randomized 1:1 to placebo or simvastatin for the next 4 wks
  Simvastatin: The study uses the Sequential Parallel Comparison design (SPCD), with two 4-week phases: Subjects are randomized 1:1 to simvastatin versus placebo add-on for 4 weeks, with the nonresponders re-randomized 1:1 for a further 4 weeks. The SPCD will allow us to pool data from both phases to estimate the simvastatin treatment effect. Subjects who respond in phase 1, and all subjects who receive simvastatin in phase 1, continue blinded treatment in phase 2 to preserve the blind, but only phase 1 results are analyzed. Dosage for simvastatin or matched placebo 20mg daily for 8 weeks.
  Placebo: Subjects are randomized to placebo add-on for 4 weeks, with the nonresponders re-randomized 1:1 to statin vs placebo for a further 4 weeks. Subjects who respond in phase 1 continue blinded treatment in phase 2 to preserve the blind, but only phase 1 results ar
- Placebo-Placebo: Placebo nonresponders for the 1st 4 weeks will be re-randomized 1:1 to placebo or simvastatin for the subsequent 4 weeks
  Placebo: Subjects are randomized to placebo add-on for 4 weeks, with the nonresponders re-randomized 1:1 to statin vs placebo for a further 4 weeks. Subjects who respond in phase 1 continue blinded treatment in phase 2 to preserve the blind, but only phase 1 results are analyzed. Dosage for simvastatin or matched placebo 20mg daily for 8 weeks.
Period: Overall Study
Arm/Group | Simvastatin-Simvastatin | Placebo->Simvastatin | Placebo-Placebo
Started | 2 | 0 | 2
Completed | 1 | 0 | 1
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin-Simvastatin | Placebo->Simvastatin | Placebo-Placebo | Total
Number analyzed (Participants) | 2 | 0 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2 | 4
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 41.5 [27 to 56] |  | 46.5 [44 to 49] | 44 [27 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 2 | 2
  Male | 2 |  | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in MADRS (4 Weeks)
Description: Change in Montgomery-Asberg Depression Rating Scale (MADRS) in simvastatin-treated epochs versus placebo-treated epochs
Time Frame: Baseline vs week 4 (and, for placebo nonresponders in 1st 4 weeks, week 8 vs week 4)
Measure: Number; unit: units on a scale
Arm/Group | Simvastatin-Simvastatin | Placebo->Simvastatin | Placebo-Placebo
Number analyzed (Participants) | 1 | 0 | 1
units on a scale | -20 |  | -10

ADVERSE EVENTS:
Arm/Group | Simvastatin-Simvastatin | Placebo->Simvastatin | Placebo-Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated early because delays in study initiation and insufficient recruitment. Our statisticians have advised us that this analysis is uninformative as it represents the change for one individual in 2 of the three arms of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No